CLINICAL TRIAL: NCT05841524
Title: Thrombus Formation Prediction in Abdominal Aneurysms Using Vector Flow Imaging
Brief Title: Vector Velocity Imaging in AAA Patients
Acronym: AAA-VFI
Status: Active, not recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); University of Twente (Other)
Responsible Party: Sponsor
Other Study IDs: 238649
Record Dates: First submitted 2023-04-12; First posted 2023-05-03 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aneurysm; Thrombus
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AAA patients, without intraluminal thrombus: patients diagnosed with an abdominal aneurysm, with a diameter below the treatment threshold of 5.5 cm and without intraluminal thrombus.
  Interventions: Diagnostic Test: Vector flow imaging measurement
- AAA patients, with intraluminal thrombus: patients diagnosed with an abdominal aneurysm, with a diameter below the treatment threshold of 5.5 cm and with intraluminal thrombus.
  Interventions: Diagnostic Test: Vector flow imaging measurement

INTERVENTIONS:
Diagnostic Test: Vector flow imaging measurement — Ultrasound measurement, using high framerate measurement techniques.

SUMMARY:
The goal of this observational study is to perform an in vivo feasibility study using real time (3D) ultrasound based vector flow imaging in 10 AAA patients (5 with intraluminal thrombus and 5 without intraluminal thrombus). Furthermore, the investigators will investigate the added value of contrast microbubbles in these high framerate, plane wave ultrasound measurements.

Included patients will undergo ultrasound scanning of their AAA, using multiple ultrasound sequences. Sequences will be tested with and without the addition of ultrasound contrast microbubbles.

DETAILED DESCRIPTION:
Currently a AAA diameter > 5.5 cm is the cut-off for treatment with the rationale that rupture risk outweighs risk of surgery at that point. Although in large cohorts such thresholds adequately reflect the repair indication, they fail in case of patient-specific decision-making. This is reflected by the fact that both small AAA rupture and large AAA's have been documented to be stable. Moreover, recently introduced biomechanical parameters show promising results with respect to improved rupture risk prediction. A key parameter is intraluminal thrombus (ILT) formation at the vessel wall, which is observed in 75% of AAA's. Recent work has shown ILT to be promoting rupture risk, outweighing its protective effect by reducing wall stress. An explanation lies in the fact that the vessel wall is primarily oxygenated due to luminal oxygen diffusion and ILT decreases oxygen supply to the AAA wall by as much as 95%. This, in turn, leads to hypoxia, inflammation and vessel wall weakening, promoting AAA rupture. Others have also shown that small AAA's (< 6 cm) that ruptured have a significantly higher volume percentage of ILT. Biomechanics behind the formation of ILT indicate that aneurysmal blood flow plays a role, in combination with the complex and patient-specific AAA geometry, inducing blood flow perturbations, e.g. vortices and stagnation zones. These local blood flow perturbations facilitate platelet adhesion and ILT formation in regions of slow and stagnant flow, in turn increasing AAA growth and the associated rupture risk. This project is a first step to quantify in vivo AAA blood flow, using high frame rate ultrasound techniques, to perform both better risk stratification and risk management.

Conventional color Doppler imaging is performed using focused ultrasound beams, which limits the achievable frame rates to approximately 25 frames per second (fps). Recent developments in computer hardware and software has enabled a shift towards unfocused imaging, where anatomical ultrasound images can be made using only a single unfocused ultrasound pulse. With the new technology, the frame rate limit is suddenly increased by a factor of 500, which results in increased flexibility when designing imaging sequences. Extremely high frame rates can now be traded for increased complexity, enabling new information to be obtained.

In this project, the investigators will use continuous, high frame rate, ECG gated, 3D slice acquisition to quantify blood flow at the inflow of the aneurysm. This will result in a vector flow imaging dataset, including the through plane component. The received signal is based on the in vivo scattering properties of blood. However, the technique might benefit from the addition of ultrasound contrast agents, therefore a second set of measurements will be obtained after intravenous injection of a contrast agent (SonoVue).

The hypothesis is that high frame rate 3D ultrasound can be used to image aneurysm blood flow. From these measurements the investigators expect that travel distance analysis shows different outcomes between AAA patients with and without intraluminal thrombus. In turn this is another piece of the puzzle to stratify patients having a higher risk of aneurysm rupture.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AAA
* AAA diameter below treatment threshold of 5.5 cm

Exclusion Criteria:

* Hypersensitivity to the active substance(s) or any of the excipients in Sonovue
* Right-to-left cardiac shunt
* Severe pulmonary hypertension (pulmonary artery pressure > 90mmHg)
* Uncontrolled systemic hypertension
* Severe pulmonary disease (e.g. COPD GOLD 3 or 4, adult respiratory distress syndrome)
* Clinically unstable cardiac disease (recent, < 3 months, or ongoing myocardial infarction, unstable angina at rest, recent percutaneous coronary intervention, clinically worsening cardiac symptoms, severe cardiac arrhythmia's, endocarditis, etc.)
* Prosthetic valves
* Loss of renal function (GFR < 31 ml/min), end-stage renal disease
* End-stage liver disease
* Sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with an AAA. Both with and without intraluminal thrombus present.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility scoring for obtaining blood flow measurements in the AAA | Through study completion, an average 6 months
  Scoring of the obtained data will be performed by a group of 5 experts

SECONDARY OUTCOMES:
Additional value of microbubble contrast injections on signal to noise ratio | Through study completion, an average 6 months
  Measurements will be performed with and without contrast, added value on signal to noise ratio will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Seternes, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olavs hospital, Trondheim University Hospital, Trondheim, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: No